CLINICAL TRIAL: NCT06372288
Title: Theta Burst Transcranial Magnetic Stimulation for the Treatment of Methamphetamine Use Disorder
Brief Title: Theta Burst TMS for Treatment of Methamphetamine Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Sooraj John, Physician, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-1754
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Methamphetamine Abuse
Keywords: Transcranial Magnetic Stimulation (TMS); methamphetamine use disorder
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either receive 5 transcranial magnetic stimulations or 5 sham transcranial magnetic stimulation (no therapeutic levels of stimulation) sessions.
Who Masked: Participant, Care Provider, Investigator
Masking Description: One study personnel not involved in participant interventions will be unblinded and will randomize participants and confirm the set up of the device for the session prior to the blinded study personnel interacting with the participant. Both the participant and the blinded study personnel will not know which group the participant will be part of throughout the study sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Transcranial Magnetic Stimulation (TMS) (Experimental): This arm receives the TMS treatments.
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham-TMS (Sham Comparator): This arm receives sham TMS treatments.
  Interventions: Device: Sham Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Transcranial Magnetic Stimulation (TMS using Intermittent theta burst stimulation (iTBS)
  Other Names: TMS; iTBS
  Arms: Transcranial Magnetic Stimulation (TMS)
Device: Sham Transcranial Magnetic Stimulation — Participants will not receive intermittent theta burst stimulation during the sham-TMS sessions
  Other Names: Sham-TMS
  Arms: Sham-TMS

SUMMARY:
This study is using Transcranial Magnetic Stimulation (TMS) to determine if interventional psychiatry treatment can help with the treatment of Methamphetamine Use Disorder. Individuals with Methamphetamine Use Disorder will receive 5 consecutive TMS treatment sessions based off of randomization. Participants will be randomized to one of two groups. TMS treatment arm or sham-TMS arm.

DETAILED DESCRIPTION:
Patients who meet criteria for the study and who agree to participate in the research study will be randomized to an arm of the study by chance (like tossing a coin). The chance of receiving TMS or sham-TMS is equal. They will be enrolled in either the TMS or sham-TMS group (both groups involve 5 TMS or sham-TMS sessions). The study doctor and the participant will not know whether they are in the TMS or sham-TMS group. The purpose of this study is to determine if TMS is a potential treatment for methamphetamine use disorder. TMS is a non-invasive technique that uses magnetic pulses to temporarily stimulate specific brain areas in awake people (without the need for surgery, anesthetic, or other invasive procedures). This study will test whether a specific type of TMS (intermittent theta burst) over the forehead can produce a reduction in things that may prompt you to want to use methamphetamines.

ELIGIBILITY:
Inclusion Criteria:

* Individuals actively struggling with Methamphetamine Use Disorder
* Must be currently enrolled in Carilion Clinic Office Based Addiction Treatment (OBAT) program

Exclusion Criteria:

- Individuals currently struggling with alcohol use and/or benzodiazepine use

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Stimulant Craving Questionnaire (STCQ) | Baseline/Visit 2, daily during iTBS/Sham-TMS, 3 days after-, 1 week after-, 2 weeks-after, and one month after completion of iTBS/Sham TMS
  Self-rated cravings for stimulants
Urine Drug Screen (UDS) | Baseline/Visit 2, day 5 of iTBS/Sham TMS, 3 days after-, 1 week after-, 2 weeks-after, and one month after completion of iTBS/Sham TMS
  Urine drug screens

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7 (GAD-7) | Screening/Visit1 and day 5 of iTBS/Sham TMS
  Self-rated anxiety severity
Patient Health Questionnaire-9 (PHQ-9) | Screening/Visit 1 and day 5 of iTBS/Sham TMS
  self-rated depression severity
Quality - Life Enjoyment Scale - Questionnaire (Q-LES-Q) | Baseline/Visit 2, day 5 of iTBS/Sham TMS, 3 days after-, 1 week after-, 2 weeks-after, and one month after completion of iTBS/Sham TMS
  Self-rated Quality of Life scale
Hamilton Anxiety Scale (HAM-A) | Baseline/Visit 2, day 5 of iTBS/Sham TMS, 3 days after-, 1 week after-, 2 weeks-after, and one month after completion of iTBS/Sham TMS
  Clinician rated anxiety
Montgomery Asberg Depression Rating Scale (MADRS) | Screening/Visit 1, Baseline/Visit 2, day 5 of iTBS/Sham TMS, 3 days after-, 1 week after-, 2 weeks-after, and one month after completion of iTBS/Sham TMS
  Clinician rated depression
Clinical Global Impression - Severity (CGI-S) | Screening/Visit 1
  Clinician rated illness severity
Clinical Global Impression - Improvement (CGI-I) | Baseline/Visit 2, day 5 of iTBS/Sham TMS, 3 days after-, 1 week after-, 2 weeks-after, and one month after completion of iTBS/Sham TMS
  Clinician rated illness improvement

CONTACTS AND LOCATIONS:
Overall Officials: Sooraj John, M.D., Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Clinic, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Su H, Chen T, Jiang H, Zhong N, Du J, Xiao K, Xu D, Song W, Zhao M. Intermittent theta burst transcranial magnetic stimulation for methamphetamine addiction: A randomized clinical trial. Eur Neuropsychopharmacol. 2020 Feb;31:158-161. doi: 10.1016/j.euroneuro.2019.12.114. Epub 2020 Jan 2. PMID 31902567
- [Background] Liu Q, Sun H, Hu Y, Wang Q, Zhao Z, Dong D, Shen Y. Intermittent Theta Burst Stimulation vs. High-Frequency Repetitive Transcranial Magnetic Stimulation in the Treatment of Methamphetamine Patients. Front Psychiatry. 2022 Apr 26;13:842947. doi: 10.3389/fpsyt.2022.842947. eCollection 2022. PMID 35558419
- [Background] Zhao D, Li Y, Liu T, Voon V, Yuan TF. Twice-Daily Theta Burst Stimulation of the Dorsolateral Prefrontal Cortex Reduces Methamphetamine Craving: A Pilot Study. Front Neurosci. 2020 Mar 25;14:208. doi: 10.3389/fnins.2020.00208. eCollection 2020. PMID 32273837
- [Background] Wang LJ, Mu LL, Ren ZX, Tang HJ, Wei YD, Wang WJ, Song PP, Zhu L, Ling Q, Gao H, Zhang L, Song X, Wei HF, Chang LX, Wei T, Wang YJ, Zhao W, Wang Y, Liu LY, Zhou YD, Zhou RD, Xu HS, Jiao DL. Predictive Role of Executive Function in the Efficacy of Intermittent Theta Burst Transcranial Magnetic Stimulation Modalities for Treating Methamphetamine Use Disorder-A Randomized Clinical Trial. Front Psychiatry. 2021 Dec 2;12:774192. doi: 10.3389/fpsyt.2021.774192. eCollection 2021. PMID 34925101
- [Background] Chen T, Su H, Wang L, Li X, Wu Q, Zhong N, Du J, Meng Y, Duan C, Zhang C, Shi W, Xu D, Song W, Zhao M, Jiang H. Modulation of Methamphetamine-Related Attention Bias by Intermittent Theta-Burst Stimulation on Left Dorsolateral Prefrontal Cortex. Front Cell Dev Biol. 2021 Aug 3;9:667476. doi: 10.3389/fcell.2021.667476. eCollection 2021. PMID 34414178
- [Background] Hanlon CA, Dowdle LT, Correia B, Mithoefer O, Kearney-Ramos T, Lench D, Griffin M, Anton RF, George MS. Left frontal pole theta burst stimulation decreases orbitofrontal and insula activity in cocaine users and alcohol users. Drug Alcohol Depend. 2017 Sep 1;178:310-317. doi: 10.1016/j.drugalcdep.2017.03.039. Epub 2017 May 30. PMID 28686990
- [Background] Su H, Zhong N, Gan H, Wang J, Han H, Chen T, Li X, Ruan X, Zhu Y, Jiang H, Zhao M. High frequency repetitive transcranial magnetic stimulation of the left dorsolateral prefrontal cortex for methamphetamine use disorders: A randomised clinical trial. Drug Alcohol Depend. 2017 Jun 1;175:84-91. doi: 10.1016/j.drugalcdep.2017.01.037. Epub 2017 Mar 29. PMID 28410525
- [Background] Cole EJ, Stimpson KH, Bentzley BS, Gulser M, Cherian K, Tischler C, Nejad R, Pankow H, Choi E, Aaron H, Espil FM, Pannu J, Xiao X, Duvio D, Solvason HB, Hawkins J, Guerra A, Jo B, Raj KS, Phillips AL, Barmak F, Bishop JH, Coetzee JP, DeBattista C, Keller J, Schatzberg AF, Sudheimer KD, Williams NR. Stanford Accelerated Intelligent Neuromodulation Therapy for Treatment-Resistant Depression. Am J Psychiatry. 2020 Aug 1;177(8):716-726. doi: 10.1176/appi.ajp.2019.19070720. Epub 2020 Apr 7. PMID 32252538